CLINICAL TRIAL: NCT03827616
Title: A Prospective Randomized Phase II Clinical Trial of Moderately Hypofractionated Radiotherapy (70 Gy in 28 Fractions vs 60 Gy in 20 Fractions) Using Helical Tomotherapy.
Brief Title: Moderately Hypofractionated Radiotherapy for Prostate Cancer.
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Tatarstan Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: prostata116
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Prostatic Neoplasms; Genital Neoplasms
Keywords: Prostate cancer; Radiation therapy; Hypofractionated radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2,5 Gy (Active Comparator): hypofractionated dosing 28 fractions x 2,5 Gy over 38 days (prostate 28 x 2,5Gy - 70Gy, seminal vesicles 28 x 2Gy - 56 Gy, node lympaticus ( if Rouch formula> 15% or N1) 28 x 1,8 Gy - 50,4 Gy).
  Interventions: Radiation: Hypofractionated IMRT using helical Tomotherapy.
- 3 Gy (Active Comparator): hypofractionated dosing 20 fractions x 3 Gy over 26day (prostate 20 x 3Gy - 60Gy, seminal vesicles 20 x 2,5Gy - 50 Gy, node lympaticus ( if if Rouch formula> 15% or N1 ) 20 x 2,2 Gy - 44 Gy).
  Interventions: Radiation: Hypofractionated IMRT using helical Tomotherapy.

INTERVENTIONS:
Radiation: Hypofractionated IMRT using helical Tomotherapy. — 70 Gy in 28 fractions intensity-modulated radiotherapy (IMRT)
  Arms: 2,5 Gy
Radiation: Hypofractionated IMRT using helical Tomotherapy. — 60 Gy in 20 fractions intensity-modulated radiotherapy (IMRT) using helical Tomotherapy.
  Arms: 3 Gy

SUMMARY:
Radiation therapy is one of the standard treatments for men with prostate cancer. Moderately hypofractionated radiotherapy has been established to be equivalent to standard fractionated radiotherapy in several large randomized clinical trials, however different hypofractionated regimens have been used in these studies. The two most common hypofractionated regimens are 70 Gy in 28 fractions and 60 Gy in 20 fractions, both are considered standard of care, however it is not unknown which regimen is better in terms of effectiveness and toxicity. The aim of this randomized controlled clinical trial is to compare the two hypofractionated radiotherapy regimens using Helical Tomotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

Compare the biochemical relapse free survival (DFS) of patients with prostate cancer treated with hypofractionated regimens 70 Gy in 28 fractions and 60 Gy in 20 fractions intensity-modulated radiotherapy (IMRT) using helical Tomotherapy.

Secondary

Compare time to local progression, freedom from biochemical recurrence, and disease-specific and overall survival of patients treated with these regimens.

Determine the incidence of gastrointestinal and genitourinary toxic effects in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to TNM ( T1-3N0M0), Gleason score (6,7 (3+4), 7(4+3), 8). Before radiotherapy patients receive hormone therapy from 3 months to 6 months. Patients are randomized to 1 of 2 treatment arms.

Arm 1 hypofractionated dosing 28 fractions x 2,5 Gy over 38 days (prostate 28 x 2,5Gy - 70Gy, seminal vesicles 28 x 2Gy - 56 Gy, node lympaticus ( if Rouch formula> 15% or N1) 28 x 1,8 Gy - 50,4 Gy).

Arm II hypofractionated dosing 20 fractions x 3 Gy over 26day (prostate 20 x 3Gy - 60Gy, seminal vesicles 20 x 2,5Gy - 50 Gy, node lympaticus ( if if Rouch formula> 15% or N1 ) 20 x 2,2 Gy - 44 Gy).

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed adenocarcinoma of the prostate. 2 The presence of the following studies: TRUS of the prostate gland, pelvis MRI, OSG.

3 Histological evaluation of prostate biopsy with assignment of the Gleason index.

4 Clinical stage T1-3N0M0 (AJCC 7th edition). 5 ECOG performance status 0-1 6 Age limit 18 years. 7 Patient consent to participate in a clinical study.

Exclusion criteria:

1. Prior or concurrent lymphomatous/hematogenous malignancy or other invasive malignancy except nonmelanomatous skin cancer or any other cancer for which the patient has been continually disease-free for ≥ 5 years (e.g., carcinoma in situ of the bladder or oral cavity)
2. Distatnt metastases.
3. Metastases in the lymph nodes of prostate cancer.
4. Radical prostatectomy or cryodestruction of the prostate gland in history.
5. Radiation of a small pelvis in the anamnesis. Bilateral orchectomy history.
6. Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months, transmural myocardial infarction within the past 6 months, acute bacterial or fungal infection requiring IV antibiotics, chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study treatment, hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical Relapse Free Survival Rate | Analysis occurs after all patients have been followed for five year.
  Determine what regime of hypofractionation will be the best 5-10 year biochemical disease free survival. Compare the results of hypofractional regimes (60Gy in 20 farctions; 70 Gy in 28 farctions).
Biochemical Relapse Free Survival Rate | Analysis occurs after all patients have been followed for ten year.
  Determine what regime of hypofractionation will be the best 5-10 year biochemical disease free survival. Compare the results of hypofractional regimes (60Gy in 20 farctions; 70 Gy in 28 farctions).

SECONDARY OUTCOMES:
Five year Local Progression Rate | Analysis occurs after all patients have been followed for five year.
  Clinical criteria for local recurrence are progression (increase in palpable abnormality) at any time, failure of regression of the palpable tumor by 2 years, and redevelopment of a palpable abnormality after complete disappearance of previous abnormalities. Histologic criteria for local recurrence are presence of prostatic carcinoma upon biopsy and positive biopsy of the palpably normal prostate more than 2 years after the start of treatment. The arms were not statistically compared because of an insufficient number of events.
Ten year Local Progression Rate | Analysis occurs after all patients have been followed for ten year.
  Clinical criteria for local recurrence are progression (increase in palpable abnormality) at any time, failure of regression of the palpable tumor by 2 years, and redevelopment of a palpable abnormality after complete disappearance of previous abnormalities. Histologic criteria for local recurrence are presence of prostatic carcinoma upon biopsy and positive biopsy of the palpably normal prostate more than 2 years after the start of treatment. The arms were not statistically compared because of an insufficient number of events.
Five year Overall Survival Rate | Analysis occurs after all patients have been followed for five year.
  Five-year rates Kaplan-Meier estimates. Overall survival (OS) was measured from study entry until the date of death. Patients still alive at the time of analysis were censored at the date of last follow-up
Ten year Overall Survival Rate | Analysis occurs after all patients have been followed for ten year.
  Five-year rates Kaplan-Meier estimates. Overall survival (OS) was measured from study entry until the date of death. Patients still alive at the time of analysis were censored at the date of last follow-up
Frequency of Patients With GU and GI Acute and Late Toxicity | Acute toxicity is measured from start of treatment to 90 days from the completion of treatment. Late toxicity is defined as toxicity occuring after 90 days from completion of treatment. Analysis occured at the time of the primary endpoint analysis.
  The frequency of GU and GI adverse events as defined and graded according to the National Cancer Institute СTCAE v4 were compared between treatment arms. Acute toxicity was defined as any toxicity beginning within 90 days of completion of RT, and late toxicity was defined as any toxicity beginning more than 90 days after the completion of RT. Acute and late GU and GI toxicity rates were tabulated and reported in two ways: dichotomized as < grade 2 vs ≥ grade 2, and dichotomized as < grade 3 vs ≥ grade 3. Higher grade indicates more severity.
Five year Quality of life measured with EQ5D. | Analysis occurs after all patients have been followed for five year.
  Compare quality of life of patients in 2 groups using the scale EQ5D (European Quality of Life Questionnaire).
Five year Quality of life measured with EPIС СP. | Analysis occurs after all patients have been followed for five year.
  Compare quality of life of patients in 2 groups using the scale EPIС СP (Expanded Prostate Cancer Index Composite for Clinical Practice).
Ten year Quality of life measured with EQ5D. | Analysis occurs after all patients have been followed for ten year.
  .Compare quality of life of patients in 2 groups using the scale EQ5D (European Quality of Life Questionnaire).
Ten year Quality of life measured with EPIС СP. | Analysis occurs after all patients have been followed for ten year.
  Compare quality of life of patients in 2 groups using the scale EPIС СP (Expanded Prostate Cancer Index Composite for Clinical Practice)

CONTACTS AND LOCATIONS:
Locations (1):
- Tatarstan Cancer Cente, Kazan', Tatarstan Republic, Russia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03827616/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03827616/ICF_001.pdf